CLINICAL TRIAL: NCT03779529
Title: EVOO-coratina Intervention on Lipids in Non-diabetic Hypertensive (h) Patients With Hyperlipidemia (h) Undergoing Periodic Hemodialysis (h)
Brief Title: EVOO Coratina Intervention on Lipids in Non-diabetic Hypertensive Patients Undergoing Hemodialysis (EVOOC-3H)
Acronym: EVOOC-3H
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Schena (Other)
Collaborators: University of Bari (Other)
Responsible Party: Principal Investigator, Francesco Paolo Schena, President and scientif director, Fondazione Schena
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2018-08-28; First posted 2018-12-19 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Chronic Kidney Disease Stage V
Keywords: olive oil; hemodialysis; lipids
MeSH Terms: interventions — Olive Oil

STUDY DESIGN:
Intervention Model Description: The general linear model for repeated measurements will be used with multiple paired comparisons in order to assess differences between the groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The olive oils will be administered as oil A or B with content unknown to participants, investigators and outcome assessors
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm label extra-vergin olive oil (EVOO) (Active Comparator): Participants will ingest two tablespoons of extra-vergin olive oil (EVOO) Coratina during the day: one spoon containing 10g of olive oil (>5mg of total biophenols/kg of olive oil) at lunch and one at dinner. The total biophenols ingested per day will be >10mg.
  Interventions: Dietary Supplement: Olive oil
- Arm label refined olive oil (ROO) (Active Comparator): Participants will ingest two tablespoons of refined olive oil during the day: one spoon containing 10 g of refined olive oil at lunch and one at dinner.
  Interventions: Dietary Supplement: Olive oil

INTERVENTIONS:
Dietary Supplement: Olive oil — Intervention includes dosage and amount of biophenols administered daily

SUMMARY:
Twenty-four non-diabetic hypertensive and hyperlipidemic patients undergoing periodic chronic hemodialysis will be enrolled for receiving extravirgin olive oil (EVOO) Coratina (12 patients) or refined olive oil (12 patients). Aim of the study is to evaluate the effect of EVOO-C on serum lipid levels. Randomization will be done centrally with appropriate stratification. Sample size is opportunistic because this is a pilot study. Dietary and clinical monitoring will be done by nephrologists, cardiologists and dieticians.

DETAILED DESCRIPTION:
Detailed Description: EXTRAVIRGIN OLIVE OIL CORATINA INTERVENTION ON LIPIDS IN NON-DIABETIC HYPERTENSIVE (H) PATIENTS WITH HYPERLIPIDEMIA (H)UNDERGOING PERIODIC HEMODIALYSIS (H) (EVOOC-3H) INTRODUCTION What is known. The primary causes of death in patients undergoing chronic hemodialysis (HD) are the cardiovascular events.

Cardiovascular risk factors(hypertension, type 2 diabetes, obesity, high levels of low density lipoprotein (LDL) , low levels of high density lipoprotein cholesterol (HDL), smoking and reduced physical activity) are almost universally present in people on HD. Evidence from randomized clinical trials demonstrate that statin administration in patients undergoing HD does not reduce the risk of adverse vascular outcomes. In the general population, there is growing evidence that the Mediterranean diet supplemented with olive oil implies cardiovascular and survival advantage. The favorable effects of the extravirgin olive oil (EVOO) are due to the combination of high content of monounsaturated fatty acids (MUFA) and polyphenols. The EVOO Coratina (EVOOC), produced in the Puglia Region within the Bari Province, is characterized by high values of polyphenols ranging between 400 and 1000 mg/kg of EVOO.

What is unknown. The potential effects of EVOOC in people on HD have not been formally explored both for surrogate and patient level endpoints.

Why this study. The investigators want to evaluate the effects of EVOOC in non-diabetic hypertensive patients undergoing chronic HD on a series of surrogate endpoints.

AIM OF THE PROPOSAL The investigators will investigate the effects of EVOOC with high content of polyphenols compared with refined olive oil (ROO) on lipid levels in HD patients.

STUDY DESIGN

Participants:

The investigators will enroll non-diabetic hypertensive and hyperlipidemic patients undergoing chronic HD Hypertension will be defined as systolic blood pressure >130 mmHg and diastolic blood pressure >80 mmHg or having any antihypertensive agents.

Hyperlipidemia will be defined as LDL cholesterol values more than 70 mg/dl or receiving statins at any dose.

Eligible patients may be of age. (40-80 years old)

The following patients will be excluded:

1. Baseline disease other than diabetic kidney disease or hypertensive kidney disease
2. Severe heart failure (NYHA class III or IV)
3. Patients with low compliance
4. Smoking, intake of antioxidant supplements (eg, carotenoids, vitamin C, vitamin E and glutathione), aspirin, or any other drug with established antioxidant properties, hyperlipidemia, obesity (body mass index >30 kg/m2), diabetes, celiac or other intestinal disease, life-threatening
5. Life expectancy <6 months based on managing physicians assessment
6. Inability to participate in the trial based on managing physician assessment

Interventions:

The experimental intervention will be EVOOC. Participants will ingest two tablespoons of olive oil during the day: one spoon containing 10g of EVOOC (>5mg of total biophenols/kg of EVOOC) at lunch and one at dinner. Total biophenols ingested per day will be >10mg.

Comparator:

The control will be refined olive oil (ROO). Participants will ingest two tablespoons of ROO during the day: one spoon containing 10g of ROO at lunch and one at dinner.

Cointerventions:

Patients may be receiving any drug for anemia, bone disease, nutrition and other including dietary advice towards a Mediterranean dietary pattern.

Patients may be on either chronic HD or hemodiafiltration (HDF). All treatments will be high flux.

CASE REPORT FORM This includes demographic findings and laboratory data at each time visit during the follow-up. Moreover, inclusion and exclusion criteria will be present at randomization time Daily food and individual quantities will be recorded on 'ad hoc' designed case report form. The intake of food will be analyzed and converted into nutrients using the useful software Medisystems (Anthropometric variable -weight) will be measured during the study.

Physical activity will be evaluated by the Minnesota Leisure Time Physical Activity Questionnaire. No restriction of physical activity will be given.

Methods:

This study will be a centrally randomized trial with blinding of participants, investigators and outcome assessors, based on the intention to treat principle.

Organizational aspects:

The study will be conducted by the Schena Foundation in collaboration with the Renal Unit at Policlinic,University of Bari, and the MED&FOOD spin-off of the University of Bari.

Follow-up duration will be 12 weeks. Clinical visit and laboratory control will be done every 4 weeks for 3 consecutive months.

Randomization:

Randomization will be performed centrally at the Schena Foundation, with appropriate stratification.

Sample size:

Sample size is opportunistic. The investigators will recruit a total of 24 individuals of whom 12 will receive EVOOC and 12 will receive ROO, based on the pilot nature of this study. There are, therefore, no formal sample size calculations.

FOLLOW- UP Dietary and clinical monitoring will be done by nephrologists, cardiologists and dieticians. Participants in both groups will receive dietary counseling. The counseling will be accompanied by written information with detailed description of typical ingested foods and the use of specific questionnaires: 1) the 14-items for the adherence to the Mediterranean diet; 2) the 137-items for the food frequency; 3) the Minnesota questionnaire for the physical activity; 4) the short-form-36 for the quality of life.

CARDIOLOGY INVESTIGATIONS

* Intima-media thickness study will be done by the measurement of the carotid-wall intima-media thickness (cIMT). Echo-measurements will be made in three zones: (a) proximal zone: about 2 cm before the flow-divider; (b) distal zone: about ½ cm before the flow-divider; (c) middle zone. These data will be used to obtain the arithmetical mean cIMT value.
* Brachial artery reactivity study will be carried out by the ultrasonographic assessment of endothelial dependent flow-mediated vasodilation of the brachial artery. ECG
* 24 hours ECG Holter monitoring
* 2D Color Doppler Echocardiography Cardiological investigations will be held during the long intradialytic period except for the ECG Holter monitoring that will be done at least one hour before and four hours after dialysis.

OUTCOMES

Outcomes will be:

* cardiovascular event onset
* composite outcome: myocardial infarction, revascularization, ischemic stroke, peripheral artery disease, cardiovascular death
* blood concentration of LDL and HDL cholesterol, total cholesterol,
* blood pressure METHODS Blood samples will be drown in the morning after 12 hours of fasting. Urine sample will be collected from the first spot morning micturition in presence of residual diuresis.

Blood and urine sample will be collected at the randomization visit and at each intervention period (every 4 weeks for a total of 3 months) after the short interval between two dialysis sessions.

Peripheral blood mononuclear cells (PBMCs) will be collected for the genome study. Serum samples will be collected for the measurement of pro-inflammatory (IL-1b, IL-6, TNFa) and anti-inflammatory (IL4, IL-10) cytokines and CRP.

A few ml of urine will be collected for tyrosol and hydroxytyrosol determinations by mass-spectrometry. In addition, other metabolites will be measured by nuclear magnetic resonance.

Oxidative stress evaluation. The investigators will evaluate at T0 and after 12 weeks ROS serum concentrations by spectrophotometric method using commercially available kit (dROMs Test Diacron). The investigators will also assess the measurement of serum 8-oxodG, a marker of oxidative DNA damage by ELISA (Trevigen). The investigators will identify the nature of ROS generated in PBMCs by the peroxide-sensitive fluorescent probe 2',7'-dichlorodihydrofluorescin diacetate (DCFH, Molecular Probes). Kinetic measurements of mitochondrial ROS generation will be evaluated by measuring the linear fluorescence increase caused by the H2O2-dependent oxidation of DCFH. NADPH-dependent superoxide generation will be measured by lucigenin-enhanced chemiluminescence methods in PBMCs isolated from HD patients. In parallel, the investigators will prepare RIPA lysates of the PBMCs and evaluate the expression of the various NADPH oxidase subunits by Western blot analysis. The antibodies for gp91phox/Nox2 or Rac1 antibodies will be furnished by Upstate/Millipore; p22phox, p47phox or p67phox will be purchased from Santa Cruz Biotechnologies. Additionally, the activity of the small GTPase Rac will be evaluated by affinity precipitation using the p21-activated kinase (PAK-1) binding domain linked to glutathione S-transferase (GST-PAK-1-PBD) on glutathione-agarose beads (Millipore/Upstate Biotech.).

STATISTICAL ANALYSIS Normality of variable distribution will be assessed by analysis of skewness and kurtosis. One-factor ANOVA and Kruskall-Wallis test will be used to analyze the differences among the two groups (case-control).

The general linear model for repeated measurements will be used with multiple paired comparisons in order to assess differences between the groups.

Linearity of values across refined OO and EVOO will be determined for testing the dose-response effect of biophenolic compounds.

Sample size and power calculations are not applicable given the pilot nature of the study with recruitment of an opportunistic sample.

Primary statistical analysis: All analyses will be carried out on an intention-to-treat basis. Statistical significance will be defined as p<0.05 for a two-sided test.

CHARACTERISTICS OF EVOOC AND ROO EVOOC: This olive oil is obtained by Coratina cultivar trees that are DNA certificated.

ROO: This olive oil used as placebo is a mixture of refined OO. Fatty acid composition and polyphenol content have been determined by gas chromatography and HPLC, respectively.

Polyphenols are undetectable in ROO. The characteristics of EVOOC and ROO (nutraceutic label) are enclosed in this protocol.

The OOs will be provided by the MED&FOOD spin-off, University of Bari.

ELIGIBILITY:
Inclusion Criteria:

* The investigators will enroll non-diabetic hypertensive and hyperlipidemic patients undergoing chronic HD
* Hypertension will be defined as having a systolic blood pressure of >130 mmHg and a diastolic blood pressure >80 mmHg or having any antihypertensive agents.
* Hyperlipidemia will be defined as having LDL cholesterol values more than 100 mg/dl or receiving statins at any dose.
* Eligible patients may be of any age.

Exclusion Criteria:

* Diabetes mellitus type 1 or 2
* Severe heart failure (NYHA class IV)
* Patients with low compliance or severe psychiatric illnesses
* Smoking, intake of antioxidant supplements (eg, carotenoids, vitamin C, vitamin E and glutathione), aspirin, or any other drug with established antioxidant properties, hyperlipidemia, obesity (body mass index >30 kg/m2), diabetes, celiac or other intestinal disease, life-threatening
* Survival expectancy <6 months based on managing physicians assessment
* Inability to participate in the trial based on managing physicians assessment

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 24 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum levels of LDL cholesterol | 1st month
  Blood measurement
Serum levels of LDL cholesterol | 2nd month
  Blood measurement
Serum levels of LDL cholesterol | 3rd month
  Blood measurement
Serum levels of HDL cholesterol, | 1st month
  Blood measurement
Serum levels of HDL cholesterol, | 2nd month
  Blood measurement
Serum levels of HDL cholesterol, | 3rd month
  Blood measurement
Serum levels of total cholesterol | 1st month
  Blood measurement
Serum levels of total cholesterol | 2nd month
  Blood measurement
Serum levels of total cholesterol | 3rd month
  Blood measurement

SECONDARY OUTCOMES:
number of participants with high blood pressure | 1st month
  Monitoring of blood pressure
number of participants with high blood pressure | 2nd month
  Monitoring of blood pressure
number of participants with high blood pressure | 3rd month
  Monitoring of blood pressure
number of participants with myocardial infarction | Measurement will be done at 1st month
  Trop-1 measurement
number of participants with myocardial infarction | Measurement will be done at 2nd month
  Trop-1 measurement
number of participants with myocardial infarction | Measurement will be done at 3rd month
  Trop-1 measurement

CONTACTS AND LOCATIONS:
Overall Officials: Francesco P Schena, MD, Principal Investigator — Fondazione Schena
Locations (1):
- Fondazione Schena, Valenzano, Bari, Italy

IPD SHARING:
Plan to Share IPD: Yes
the IPD are shared with other researchers
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2 years
Access Criteria: publications or reports
URL: http://www.fondazioneschena.org

REFERENCES:
- [Background] Palmer SC, Craig JC, Navaneethan SD, Tonelli M, Pellegrini F, Strippoli GF. Benefits and harms of statin therapy for persons with chronic kidney disease: a systematic review and meta-analysis. Ann Intern Med. 2012 Aug 21;157(4):263-75. doi: 10.7326/0003-4819-157-4-201208210-00007. PMID 22910937
- [Background] Estruch R, Martinez-Gonzalez MA, Corella D, Salas-Salvado J, Ruiz-Gutierrez V, Covas MI, Fiol M, Gomez-Gracia E, Lopez-Sabater MC, Vinyoles E, Aros F, Conde M, Lahoz C, Lapetra J, Saez G, Ros E; PREDIMED Study Investigators. Effects of a Mediterranean-style diet on cardiovascular risk factors: a randomized trial. Ann Intern Med. 2006 Jul 4;145(1):1-11. doi: 10.7326/0003-4819-145-1-200607040-00004. PMID 16818923
- [Background] Estruch R, Ros E, Salas-Salvado J, Covas MI, Corella D, Aros F, Gomez-Gracia E, Ruiz-Gutierrez V, Fiol M, Lapetra J, Lamuela-Raventos RM, Serra-Majem L, Pinto X, Basora J, Munoz MA, Sorli JV, Martinez JA, Martinez-Gonzalez MA. Retraction and Republication: Primary Prevention of Cardiovascular Disease with a Mediterranean Diet. N Engl J Med 2013;368:1279-90. N Engl J Med. 2018 Jun 21;378(25):2441-2442. doi: 10.1056/NEJMc1806491. Epub 2018 Jun 13. No abstract available. PMID 29897867